CLINICAL TRIAL: NCT06809829
Title: Clinical and Radiographic Evaluation of Doxycycline and Doxycycline Loaded Nanoparticles With Gelatin Sponge on Immediate Implant Placement in Esthetic Zone: A Randomized Clinical Trial
Brief Title: Evaluation of Doxycycline Nanoparticle With Gelatin Sponge on Immediate Implant in Esthetic Region
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kafrelsheikh University (Other)
Responsible Party: Principal Investigator, Ahmed Othman Fathy Othman El-Kersh, demonstrator of Department of Periodontology, Oral Diagnosis and Oral Radiology at Faculty of Dentistry, Kafrelsheikh university, Kafrelsheikh University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KFSIRB200-482
Record Dates: First submitted 2025-01-30; First posted 2025-02-05 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-01

CONDITIONS: Immediate Implant Placement
Keywords: Immediate Implant Placement; Nanoparticles; Doxycycline; Gelatin Sponge

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- immediate implant placement with doxycycline loaded gelatin nano particles and gelatin sponge (Experimental)
  Interventions: Procedure: Immediate Implant Placement
- Immediate Implant Placement with Doxycyline and Gelatin Sponge (Active Comparator)
  Interventions: Procedure: Immediate Implant Placement

INTERVENTIONS:
Procedure: Immediate Implant Placement — Eight patients undergoing immediate implant placement with the buccal gap filled with doxycycline loaded gelatin nanoparticles along with gelatin sponge (group A) Eight patients undergoing immediate implant placement with the buccal gap filled with doxycycline along with gelatin sponge (group B)

SUMMARY:
The goal of this clinical trial is to Evaluate the effect of Doxycycline nanoparticles along with gelatin sponge in immediate implant cases in esthetic zone. The main question it aims to answer is:

Does the application of doxycycline nanoparticles with gelatin sponge improve the clinical and radiographic outcomes of immediate implant cases in esthetic zone?

Researchers will compare eight patients undergoing immediate implant placement with the buccal gap filled with doxycycline loaded gelatin nanoparticles along with gelatin sponge (group A) with eight patients undergoing immediate implant placement with the buccal gap filled with doxycycline along with gelatin sponge (group B). to see if the doxycycline loaded nanoparticles will improve the clinical and radiographic outcomes of the immediate implant .

Participants will [describe the main tasks participants will be asked to do, interventions they'll be given and use bullets if it is more than 2 items].

ELIGIBILITY:
Inclusion Criteria:

* The presence of non-restorable single-rooted maxillary centrals, canines or premolars.
* Sufficient bone volume.
* Good oral hygiene.
* The remaining space between the socket and the fixture equals or more than 2mm at the coronal third of the socket.
* Sufficient bone width (≥ 1 mm) in the buccal plate of the remaining bone to place an implant confirmed by cone beam computer tomography (CBCT).

Exclusion Criteria:

* Insufficient bone volume.
* Active infection.
* Patients on chemotherapy or radiotherapy.
* Patients who have systemic disorders {uncontrolled diabetes mellitus, autoimmune disease, …etc},
* Pregnant patients,
* Patients with bone diseases
* Presence of periapical pathology affecting the neighbouring teeth.
* Smokers.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 16 (Estimated)
Dates: Start 2025-02 (Estimated); Primary Completion 2026-07 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Marginal (crestal) bone loss (MBL). | after surgery and 6 months after surgery
  Radiographic examination of the patients will be done firstly pre-operative then just after the surgical procedures as a base point and at six months follow-up period post-operative by using CBCT (carestream 9600). On Demand3D program will be used for image reconstruction and analysis. For the calculation of marginal (crestal) bone loss (MBL), the implant will be used as a reference by adjusting the cross-sectional long axis in the center of the implant and bisecting it. A line will be drawn parallel to the implant, starting at the crest of the bony cortical plate of bone and ending at the apical level of the implant; height will be recorded in millimeters immediately and 6 months postoperative. The same process will be repeated from the palatal direction.

SECONDARY OUTCOMES:
Pink Esthetic Score | before the surgery, 3 months and 6 months after the surgery
  The patients will be photographed to measure the pink esthetic sore before the surgery, 3 months, and 6 months after the surgery.
Peri-Implant Periodontal Probing depth (PPD): | 3 months and 6 months after the surgery
  This index depends mainly on the usage of 0.5 mm Michigan O probe with graduations. Measurements will be evaluated at six sites per implant i.e., the disto-facial surface, mid facial surface, mesio-facial surface, mesio-lingual surface, mid lingual surface and disto-lingual surfaces of the implant. PPD will be measured by taking the reading from the free gingival margin to the base of the pocket. The mean score of the implant will be obtained by adding the six scores and dividing it by six. Measurements will be recorded to the nearest 0.5 mm six months after implant placement (prosthetic phase) and three months after the prosthesis placement.
Peri-implant vertical bone level. | after surgery and 6 months after surgery
  Measurement will be carried out on four aspects (mesial, distal, buccal and lingual) around all implants of the selected OPGs using CBCT (carestream 9600). On Demand3D program will be used for image reconstruction and analysis. The implant shoulder and the bone ridge will be used as reference points. The distance between the implant shoulder and the bone crest directly in contact with the implant will be measured with the ruler function. The presence of peri-implant bone defect will be determined by the percent of bone loss related to the length of the implant.
Implant stability | at the time of surgery, 3 months and 6 months post surgery
  The transducer of the RFA device (Osstell®. Osstell, Baltimore) will be placed by hand tightening onto implant fixture. The implant stability quotient (ISQ) values will be measured both parallel and perpendicular to alveolar ridge of the jaw. The final ISQ value for each implant will be the mean of ISQ values. ISQ values will be measured again at re-entry after 3, 6 months for each implant.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of dentistry kafrelsheikh university, Kafrelsheikh, Kafrelsheikh, Egypt